CLINICAL TRIAL: NCT06702098
Title: Single-center and Single-arm Clinical Study of INK Cell Therapy for Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: Induced Pluripotent Stem Cells Derived Natural Killer Cells Therapy for Refractory and Relaps Acute Myelogenous Leukemia
Acronym: iNK-r/r AML
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Ruixin Biotechnological Co., LTD (Industry)
Collaborators: Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ruixin Biotech
Record Dates: First submitted 2024-11-17; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: iNK cells; R/R AML; iPSCs
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cell therapy group (Experimental): Intravenous infusion of iNK cells is given to the subject, 5*108 to 1*109 cells/dose, two doses per week, a total of 8 doses. And then 1*109 cells/dose, one doses every 4 weeks , a total of 5 doses.
  Interventions: Drug: iNK cells

INTERVENTIONS:
Drug: iNK cells — Induced pluripotent stem cells derived NK cells.

SUMMARY:
This is a clinical study on the use of iNK cells for the treatment of refractory relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
Natural killer (NK) cells are lymphocytes of the innate immune system and could recognize and kill a wide range of cells in distress, particularly tumour cells and cells infected with viruses. Induced pluripotent setm cells(iPSCs) derived NK cells have better proliferative capacity and homogeneity than donor peripheral blood or umbilical cord blood derived NK cells. We conduct this clinical study to evaluate the efficacy and safety of INK cells in the treatment of acute myeloid leukemia and our purpose is to find new treatment option.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy the following criteria to be enrolled in the study.

1. Patient is ≥ 18 and ≤ 80 years of age at the time of signing the Study informed consent form (ICF).
2. Patient understands and voluntarily signs the Study ICF prior to any study-related assessments/procedures are conducted.
3. Patient has eligible disease status:

   3.1 Primary or Secondary acute myeloid leukemia (AML) Patients in first of second Morphological Complete Remission (CR), Morphological Complete Remission with incomplete hematologic recovery (CRi), or Morphologic Leukemia-free State (MLFS) as defined by the European LeukemiaNet (ELN) recommendations for AML Response Criteria (Dohner, 2017).

   3.2 R/R diagnosis based on confirmed diagnosis with local pathology report following any reinduction/ salvage therapy ELN guidelines.

   3.2.1 Relapsed AML are defined as having relapsed after achieving ≥ 1 CR, including relapse after allogeneic stem cell transplantation (≥ 2 months after transplant).

   3.2.2 Refractory AML, defined as not achieving CR, CRi, or MLFS after 2 or more cycles of induction therapy (primary refractory) or not achieving CR after treatment for relapsed AML.

   3.2.3 Secondary AML (MDS transformation): Secondary AML patients are eligible to participate if they have received a minimum of one prior line of treatment for AML.

   3.2.4 Treatment-related AML: Treatment-related AML patients are eligible to participate if they have received a minimum of one prior line of treatment for AML.
4. No active infection.
5. No heart , liver and kidney functioninsufficiency.
6. No central nervous system leukemia.

Exclusion Criteria:

1. Subject meets one of the following criteria. 1.1History of CAR-T treatment with third degree CRS. 1.2 History of NK cell and CIK cell immunotherapy.
2. Serious cardiovascular and cerebrovascular diseases. 2.1 Severe heart rhythm or conduction abnormalities, corrected QT interval (QTc)≥480 ms.

   2.2 Complete left bundle branch block, second- or third-degree atrioventricular block; 2.3 Severe, uncontrolled cardiac arrhythmias requiring medication. 2.4 New York Heart Association (NYHA) class II or above congestive heart failure.

   2.5 Left ventricular ejection fraction (LVEF) <50% in color Doppler echocardiography.

   2.6 History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, severe pericardial disease, ECG evidence of acute ischemic or active conduction system abnormalities within 6 months prior to recruitment.
3. Previous or present concomitant other malignancies (except for basal cell carcinoma of the skin, non-melanoma and non-melanoma, carcinoma in situ of the breast/cervix that have been effectively controlled, and other malignancies that have been effectively controlled without treatment in the past five years).
4. Uncontrollable systemic disease(e.g. uncontrolled hypertension, diabetes, etc).
5. Pregnant women, lactating females, patients who refuse to use effective contraception during the study.
6. history of severe neurological or psychiatric illness.
7. Positive for hepatitis B surface antigen.
8. Patients who are judged by the investigator to be unsuitable for participating in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
MRD negative rate | 12 months
Progression-free Survival | 12 months
Overall survival | 12 months

SECONDARY OUTCOMES:
Determination of chimerism of iNK cells in peripheral blood of subject. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Huo Tan, MD, Principal Investigator — Fifth Affiliated Hospital of Guangzhou Medical University; Runhui Zheng, MD, Study Director — Fifth Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou Ruixin Biotechnology Co., Ltd, Guangzhou, Guangdong Province, China, China

IPD SHARING:
Plan to Share IPD: Yes
What data in particular will be shared? Individual participant data that underlie the results reported in this article, after deidenti- fication (text, tables, figures, and appendices).
  What other documents will be available？ Study Protocol. When will data be available (start and end dates)? Beginning 9 months and ending 36 months following article publication. With whom? Investigators whose proposed use of the data has been approved by an independent review committee(learned intermediary) identified for this purpose.
  For what types of analyses? For individual participant data meta-analysis. By what mechanism will data be made available? Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in clinical research center of the fifth affiliated hospital of Guangzhou medical university (https://www.gyfwyy.com/gcp/).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee(learned intermediary) identified for this purpose.
URL: https://www.gyfwyy.com/gcp/